CLINICAL TRIAL: NCT00830076
Title: A Study to Assess the Effects of Co-Administration of Sitagliptin and Metformin on Incretin Hormone Concentrations
Brief Title: A Study of the Effects of Co-Administration of Sitagliptin (MK-0431) and Metformin on Incretin Hormone Concentrations (MK-0431-110)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-110; 2009_521
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sitagliptin + placebo metformin (Experimental)
  Interventions: Drug: sitagliptin phosphate; Drug: Comparator: placebo metformin
- Metformin + placebo sitagliptin (Experimental)
  Interventions: Drug: metformin hydrochloride; Drug: Comparator: placebo sitagliptin
- Sitagliptin + metformin (Experimental): Co-administration of sitagliptin and metformin
  Interventions: Drug: sitagliptin phosphate; Drug: metformin hydrochloride
- Placebo sitagliptin + placebo metformin (Placebo Comparator): Co-administration of placebo to sitagliptin and placebo to metformin
  Interventions: Drug: Comparator: placebo sitagliptin; Drug: Comparator: placebo metformin

INTERVENTIONS:
Drug: sitagliptin phosphate — Sitagliptin 100 mg tablet on Day 1 and Day 2 in the morning. There will be a 7-day washout between treatment periods.
  Other Names: Januvia
  Arms: Sitagliptin + metformin; Sitagliptin + placebo metformin
Drug: metformin hydrochloride — Metformin 500 mg tablet in the morning and evening on Day 1 and two 500 mg tablets of metformin (total dose 1000 mg) on Day 2 in the morning. There will be a 7-day washout between treatment periods.
  Other Names: Glucophage
  Arms: Metformin + placebo sitagliptin; Sitagliptin + metformin
Drug: Comparator: placebo sitagliptin — Placebo to sitagliptin 100 mg in the morning on Days 1 and 2. There will be a 7-day washout between treatment periods.
  Arms: Metformin + placebo sitagliptin; Placebo sitagliptin + placebo metformin
Drug: Comparator: placebo metformin — Placebo to metformin 500 mg tablet in the morning and evening on Day 1 and two placebo to metformin 500 mg tablets (1000 mg total dose) in the morning of Day 2. There will be a 7-day wash out between treatment periods.
  Arms: Placebo sitagliptin + placebo metformin; Sitagliptin + placebo metformin

SUMMARY:
This study will assess the effects of sitagliptin and metformin alone and after co-administration on incretin hormone concentrations in patients with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must have a negative pregnancy test
* Subject has type 2 diabetes and is not currently receiving treatment with an oral AHA agent, has not received such treatment for 3 months prior to study, and/or has not received more than 4 total weeks treatment with an oral AHA agent for 12 to 18 months prior to the study
* Subject is a nonsmoker or has not smoked and/or used nicotine for at least 6 months

Exclusion Criteria:

* Subject has a history of stroke, seizures, or major neurological disorders
* Female subject is breastfeeding
* Subject cannot refrain from use of any prescription or non-prescription drugs beginning 2 weeks prior to first dose of study drug
* Subject consumes more than 3 alcoholic beverages per day
* Subject consumes more than 6 caffeinated beverages per day
* Subject has had major surgery, or has donated or lost 1 unit of blood within 4 weeks of screening
* Subject has a history of cancer, except certain skin or cervical cancer or other cancers treated more than 10 years prior to screening
* Subject has a history of multiple and/or severe allergies or intolerance to drugs or food

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12-02 (Actual); Primary Completion 2009-04-30 (Actual); Study Completion 2009-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants received four 2-day treatment regimens (sitagliptin + placebo metformin for 2 days, metformin + placebo sitagliptin for 2 days, co-administration of sitagliptin + metformin for 2 days, and placebo sitagliptin + placebo metformin for 2 days) with a 7-day washout between each treatment period.
Period: Sitagliptin + Placebo Metformin
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0
Period: 7-day Washout
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0
Period: Metformin + Placebo Sitagliptin
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0
Period: 7-day Washout
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0
Period: Sitagliptin + Metformin
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0
Period: 7-day Washout
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0
Period: Placebo Sitagliptin + Placebo Metformin
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Incremental Post-prandial 4-hour Weighted Mean Active Glucagon-like Peptide-1 (GLP-1) Plasma Concentrations
Description: Meal was given 2 hours postdose. Blood samples for determination of active GLP-1 concentration were collected (4 hours postmeal) on Day 2 in each treatment period.
Time Frame: 6 hours postdose (4 hours postmeal) on Day 2
Measure: Least Squares Mean (95% Confidence Interval); unit: picomolar
Arm/Group | All Participants
Number analyzed (Participants) | 18
picomolar
  Sitagliptin + placebo metformin | 6.00 [4.53 to 7.94]
  Metformin + placebo sitagliptin | 4.09 [3.09 to 5.42]
  Sitagliptin + metformin | 7.22 [5.45 to 9.55]
  Placebo sitagliptin + placebo metformin | 1.55 [1.17 to 2.05]

2. Secondary Outcome: β-cell Sensitivity
Description: β-cell sensitivity was defined as the incremental post-prandial
  4-hour area under the curve (AUC) for insulin secretion rate (ISR) normalized by the incremental post-prandial 4-hour plasma glucose AUC.
Time Frame: 6 hour post-dose (4 hour postmeal) on Day 2
Population: Beta-cell sensitivity was not calculated for 1 participant following the administration of sitagliptin alone and metformin alone due to missing insulin data.
Measure: Least Squares Mean (95% Confidence Interval); unit: (ng/min)/(mg/dL)*10^ -3
Arm/Group | All Participants
Number analyzed (Participants) | 18
(ng/min)/(mg/dL)*10^ -3
  Sitagliptin + placebo metformin, n=17 | 19.50 [11.89 to 32.00]
  Metformin + placebo sitagliptin, n=17 | 25.71 [15.67 to 42.18]
  Sitagliptin + metformin, n=18 | 26.39 [16.18 to 43.05]
  Placebo sitagliptin + placebo metformin, n=18 | 15.44 [9.46 to 25.19]

3. Secondary Outcome: Incremental Post-prandial 4-hour Weighted Mean Plasma Glucose Concentrations
Description: Meal was given 2 hours postdose. Blood samples for determination of glucose concentration were collected (4 hours postmeal) on Day 2 in each treatment period.
Time Frame: 6 hours postdose (4 hours postmeal) on Day 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 18
mg/dL
  Sitagliptin + placebo metformin | 42.30 [30.51 to 54.08]
  Metformin + placebo sitagliptin | 29.33 [17.55 to 41.12]
  Sitagliptin + metformin | 20.02 [8.24 to 31.81]
  Placebo sitagliptin + placebo metformin | 51.02 [39.24 to 62.81]

ADVERSE EVENTS:
Time Frame: 43 days (four 2-day treatment periods, a 7-day washout interval between each treatment period, and approximately 14 days following the last dose of study treatment)
Groups:
- Sitagliptin + Placebo Metformin: Participants received sitagliptin + placebo metformin for 2 days.
- Metformin + Placebo Sitagliptin: Participants received metformin + placebo sitagliptin for 2 days.
- Sitagliptin + Metformin: Participants received co-administration of sitagliptin + metformin for 2 days.
- Placebo Sitagliptin + Placebo Metformin: Participants received placebo sitagliptin + placebo metformin for 2 days.
Arm/Group | Sitagliptin + Placebo Metformin | Metformin + Placebo Sitagliptin | Sitagliptin + Metformin | Placebo Sitagliptin + Placebo Metformin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4/18 | 3/18 | 3/18 | 4/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin + Placebo Metformin (N=18) | Metformin + Placebo Sitagliptin (N=18) | Sitagliptin + Metformin (N=18) | Placebo Sitagliptin + Placebo Metformin (N=18)
Iron Deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.